CLINICAL TRIAL: NCT01546662
Title: A Randomized Double Dummy Double Blind Dose Determining Place-bo Controlled Study to Evaluate Efficacy of Investigational Product E-RH-06 at 2 Dose Levels for the Metabolic Management of Chronic or Recurrent, Non-infective Nasal Congestion With-or-without Rhinorrhea.
Acronym: EB-RH-02-11
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EB-RH-02-11; EB-ERH-02-11 (Other: Self)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- E-RH-06 - Low Dose (Experimental): 1 Capsule twice daily
  Interventions: Dietary Supplement: E-RH-06
- E-RH-06 - High Dose (Experimental): 2 capsules twice daily
  Interventions: Dietary Supplement: E-RH-06
- Placebo ; (Placebo Comparator): Placebo Comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: E-RH-06 — Capsules, 1 capsule/ 2 capsule, twice daily for 12 weeks
  Other Names: Olfaclear
  Arms: E-RH-06 - High Dose; E-RH-06 - Low Dose
Dietary Supplement: Placebo — 1/ 2 capsules, twice daily for 12 weeks
  Arms: Placebo ;

SUMMARY:
The study will be conducted in two phases. First phase will be 16 weeks study to assess the safety, efficacy & to determine the most appropriate dose. Will consist of following visits.

Phase II (Extended Follow-up): At the end of Day 112, an interim analysis will be conducted to assess the sustained efficacy of the investigational product and accordingly the study will enter into phase II.

DETAILED DESCRIPTION:
The study will be conducted in two phases. First phase will be 16 weeks study to assess the safety, efficacy & to determine the most appropriate dose. Will consist of following visits:

Screening I (Day -14) Visit: After obtaining written informed consent, subjects will be screened for study eligibility as per the inclusion/exclusion criteria defined in the study protocol on screening visit. The screening evaluations will include general examination, medical history taking, recording of vital parameters and assessment of frequency of symptoms, and Total Nasal Symptom Score (TNSS) calculation. Blood sample will be collected for CBC, SGPT & Urine creatinine analysis. Simultaneously urine samples will be collected for urine routine & UPT analysis. ECG will be performed.

Screening II (Day -7) Visit: Laboratory results and ECG reports will be analysed by the investigator. Eligible subjects will be entered into 7 days run-in period. Rescue medication will be dispensed.

Baseline Visit/ Randomization Visit (Week 0): At the end of screening period (Baseline visit, window period + 3 days), subjects fulfilling the rhinitis frequency and symptom criteria (baseline average scores as: average 24-h TNSS 10 over 15 days, and requiring no more than 2 tablets of rescue medication (Loratidine) daily to control the symptoms) will be randomized to one of the 3 treatment groups to receive the following treatment regimens:

1. Group 1: E-RH-06/ 1 BID: (E-RH-06 + Placebo) Twice Daily
2. Group 2: E-RH-06/ 2 BID: (E-RH-06 + E-RH-06) Twice Daily
3. Group 3: Placebo: (Placebo + Placebo) Twice Daily Rescue medication accountability & dispensing will be performed. Specially designed rescue medication charts will be dispensed. Subjects will be provided with subject diaries. Vitals & general examination will be performed. TNS scoring will be performed. IP/ Placebo will be dispensed. IP accountability will be performed. Adverse event & serious adverse event monitoring will be performed.

Days 14 (window period plus/ minus 3 days) (Follow Up I Visit): This visit will involve general examination & vital signs recording. The frequency and intensity of symptoms as well as AE/SAE will be monitored and documented. IP/ placebo accountability & dispensing will be conducted. Rescue medication accountability & dispensing will be done. TNS scoring will be performed.

Day 28 (window period plus/ minus 3 days) (Follow Up II Visit): General examination, vital signs (Blood Pressure and Pulse) recording, documenting frequency and intensity of symptoms, monitoring of AE/SAE will be done. IP/ Placebo & rescue medication accountability & dispensing will be done. Subject diary will be assessed.

Day 56 (window period plus/ minus 3 days) (Follow Up III Visit): The visit will involve general examination & vital signs recording, documenting of frequency and intensity of symptoms, monitoring of AE/SAE and use of rescue medication. IP/ Placebo accountability & dispensing will be performed. Rescue medication will be dispensed for further usage. TNS scoring will be done.

Day 84 (window period plus/ minus 3 days) (End-of-Treatment Visit): General examination, vital signs recording, documenting frequency and intensity of symptoms, monitoring of AE/SAE will be performed. Dispensed IP/ Placebo & rescue medication will be accounted in coordination with the left medication count, rescue medication chart & patients history. TNS scoring will be performed. Placebo will be dispensed. Rescue medication will be dispensed to continue further. Blood sample will be collected for CBC, SGPT & Serum Creatinine analysis. ECG will be performed.

Day 112 (window period plus/ minus 3 days) (Post Treatment Follow Up Visit): The visit will involve general examination, vital signs recording, documenting frequency and intensity of symptoms, monitoring of AE/SAE and use of rescue medication. Rescue medication accountability will be performed. TNS scoring will be performed.

In between the follow up clinic visits, weekly scores for intensity of rhinitis symptoms will be obtained through subject diaries /telephonic assessments made at each week.

Telephonic Follow Up: Telephonic follow up will be done on Day 42, 78 & 90 to assess the nasal symptoms.

Phase II (Extended Follow-up): At the end of Day 112, an interim analysis will be conducted to assess the sustained efficacy of the investigational product and accordingly the study will enter into phase II. In case of more than/ equal to 75% subjects from individual active groups demonstrating significant sustained efficacy at week 16, the study will enter in to an open label, exploratory, extended follow-up phase for next 36 weeks (total 52 weeks). This extended follow-up phase will be conducted to determine if 12-week treatment with E-RH-06 help to reduce risk of seasonal nasal congestion with-or-without rhinorrhea during the extended follow-up period of 52-weeks. No other efficacy or safety evaluations will be carried out during this phase (extended follow-up).

ELIGIBILITY:
Inclusion Criteria:• Male and female subjects in the age group of 18-60 years with per-sistent or recurrent nasal congestion and/ or rhinorrhea as defined by the symptoms that last for not less than an hour.

* Demonstrating baseline average 24 hour TNSS ≥10.
* No clinical evidence of infection indicated by mucopurulent or puru-lent discharge, fever, and tenderness over paranasal sinuses.
* Subjects who will be able to read and fill-up subject diary efficiently.
* Able and willing to give informed consent.
* Able and willing to follow all study related instructions and to make all required visits.

Exclusion Criteria:• Subjects who have taken systemic, topical corticosteroids, long acting antihistamines or immunosuppressive medication within last 4 weeks or planning to take them within the course of the study.

* Acute febrile illness (such as cold, flu etc.) within one week of enroll-ment.
* Subjects with nasal structure deformities, nasal polyps, severe deviat-ed nasal septum and hypertrophic rhinitis will be excluded from the study.
* Clinical history of allergy/ hypersensitivity to one or more products of herbal origin.
* Pregnant / lactating women and women who are planning to get preg-nant
* Recent (within last 3 months) participation in a clinical trial
* Recent (within last 15 days) use of any herbal product for the indication under study
* Patients with severe conditions of chronic sinusitis deviated nasal sep-tum or nasal polyposis.
* Bronchial asthma patients on loading/ maintenance therapy of theophy-line.
* Patients requiring continuous use of laxatives.
* Major chronic disease of liver, kidney, CVS or CNS and other body systems
* A psychiatric condition or chronic alcohol or drug abuse problem, determined from the patient's medical history, which in the Investigator's opinion may pose a threat to patient compliance.
* Subjects otherwise judged by the investigator or sub -investigator to be inappropriate for inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
TNSS Score | 12 weeks
  To determine if the investigational product E-RH-06 relieves the symptoms of nasal congestion with-or-without rhinorrhea to a greater extent than placebo with 12 weeks' treatment as assessed by the pre-visit 24 hours reflective TNSS

SECONDARY OUTCOMES:
Reduction of frequency | 4 weeks
  Reduction in TNSS at the end of 4 weeks as compared to baseline Reduction in Total Symptom Score (TSS) and/or Total Non Nasal Symptom Score (TNNSS) at the end of 4 weeks as compared to baseline Reduction in frequency of AR attacks at the end of 4 weeks as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shalini Shrivastava, M.D, Study Chair — Enovate Biolife Pvt Ltd
Locations (4):
- India (4):
  - Shree sidhi clinic, Mumbai, Maharashtra
  - The Clinic, Mumbai, Maharashtra
  - Chirayu Clinic, Nashik, Maharashtra
  - Suyog Hospital, Nashik, Maharashtra